CLINICAL TRIAL: NCT03285412
Title: Phase II Study of CDK 4/6 Inhibitor, LEE011 (Ribociclib), in Combination With Adjuvant Endocrine Therapy at Varying Duration for ER-positive Breast Cancer (LEADER).
Brief Title: CDK 4/6 Inhibitor, Ribociclib, With Adjuvant Endocrine Therapy for ER-positive Breast Cancer
Acronym: LEADER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Arielle Janine Medford, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-232
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ribociclib + Endocrine Rx (Experimental): Ribociclib will be administered. Endocrine therapy will be administered.
  Interventions: Drug: Ribociclib; Other: Endocrine therapy
- Endocrine Rx (Active Comparator): Endocrine therapy will be administered.
  Interventions: Other: Endocrine therapy

INTERVENTIONS:
Drug: Ribociclib — Ribociclib is a drug designed to block certain proteins called cyclin-dependent protein kinases 4 and 6 (CDK4/6). These proteins are needed for cells to divide and may also control the ability of certain cancers to grow.
  Other Names: Kisqali
  Arms: Ribociclib + Endocrine Rx
Other: Endocrine therapy — Hormone therapy

SUMMARY:
This research study is studying a drug as a possible treatment for ER-positive Breast Cancer

The drug involved in this study is:

-Ribociclib

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

This research study is a study with endocrine therapy and CDK 4/6 inhibitor (ribociclib) for early breast cancer. There is no placebo in this study. The study has two components - pre-screening with ctDNA to detect minimal residual disease (pre-screening), and treatment with ribociclib in combination with endocrine therapy (main portion).

The FDA (the U.S. Food and Drug Administration) has approved ribociclib in combination with aromatase inhibitors as a treatment option for advanced/metastatic (stage IV) breast cancer.

In this research study, the investigators are evaluating efficacy of ribociclib in patients who have MRD based on ctDNA.

Ribociclib is a drug designed to block certain proteins called cyclin-dependent protein kinases 4 and 6 (CDK4/6). These proteins are needed for cells to divide and may also control the ability of certain cancers to grow. The investigators believe that ribociclib may stop the participant cancer cells from growing and dividing by blocking these CDK4/6 proteins.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have biopsy proven localized ER+ (≥ 10%), HER2 negative, invasive breast cancer, with pathological stage (including post-neoadjuvant therapy) T1c-T4c, any N, M0, by AJCC 7th edition staging. Invasive breast cancer must be ER+ in ≥10% of the cells and HER2 negative (IHC 0 or 1+ and/or FISH negative with a ratio <2) by ASCO/CAP guidelines. For IHC 2+, the tumor must be FISH negative with a ratio <2. PR status must be performed. ER, PR and HER2 measurements should be performed according to institutional (local) guidelines, in a CLIA-approved setting. Evaluation for metastatic disease is not required in the absence of symptoms. Patients must have completed definitive surgery for breast cancer.
* Detectable ctDNA
* No prior history of other malignancies within past 5 year (besides breast cancer as per 3.1.1). Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: ductal carcinoma in situ of the breast, cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin. No concurrent malignancy or other serious medical condition as deemed by the investigator.
* Participants may or may not have received (neo)adjuvant chemotherapy, but must be at least 4 weeks after last dose of chemotherapy and/or biological therapy at the time of screening, with no more than grade 1 residual toxicity (except ≤ grade 2 neuropathy or ≤ grade 2 alopecia).
* Participants may or may not have received adjuvant radiotherapy, but must be at least 30 days after last dose radiotherapy, with no more than grade 1 residual toxicity at the time of screening.
* Pre- and postmenopausal women are eligible. Premenopausal women must have a negative serum or urine pregnancy test. Pregnancy testing does not need to be pursued in female patients who are: age ≥ 60 years; or age < 60 with intact uterus and amenorrhea for 12 consecutive months or more AND estrogen (estradiol) levels within postmenopausal range; or status-post bilateral oophorectomy, total hysterectomy, or bilateral tubal ligation.
* QTc (Fredericia's formula) < 470ms.
* Must be ≥ 18 years of age.
* Prior CDK 4/6 inhibitor is permitted provided it was more than 12 months ago (from consent date).
* ECOG performance status 0-1 (Karnofsky ≥70%, see Appendix A)
* Patients may enroll within 20 years of breast cancer diagnosis, as long as there is a plan for at least 1 more year of adjuvant endocrine therapy.
* Ability to understand and the willingness to sign a written informed consent document. Patient must sign the Informed Consent (ICF) prior to any screening procedures being performed and is able to comply with protocol requirements.
* Currently on adjuvant endocrine therapy (tamoxifen and/or aromatase inhibitor (AI)), i.e prior use of any AI, including letrozole, anastrozole or exemestane, or tamoxifen is allowed. However, tamoxifen use is not allowed during the study with ribociclib. Patients on tamoxifen interested in this trial could be switched to AI on C1D1 or before/during screening. Concurrent GNRH agonist is allowed, and is recommended with AI in pre/peri-menopausal patients.
* Patient has adequate bone marrow and organ function as defined by the following laboratory values at screening:

  * Absolute neutrophil count ≥1.5 × 109/L
  * Platelets ≥100 × 109/L
  * Hemoglobin ≥9.0 g/dL
  * Potassium, total calcium (corrected for serum albumin), magnesium, sodium and phosphorus within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication
  * Serum creatinine <1.5 mg/dL or creatinine clearance ≥50 mL/min
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 x ULN.
  * Total bilirubin < ULN; or total bilirubin ≤3.0 x ULN or direct bilirubin ≤1.5 x ULN in patients with well-documented Gilbert's Syndrome.
  * Fasting plasma glucose <140 mg/dL / 7.7 mmol/L..

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants who are receiving any other investigational agents.
* Participants with known brain metastases, or any other metastases from cancer.
* Participants receiving any medications or substances that are inhibitors or inducers of CYP3A4 are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality including any of the following:

  * History of angina pectoris, symptomatic pericarditis, coronary artery bypass graft (CABG) or myocardial infarction within 6 months prior to study entry.
  * Documented cardiomyopathy.
  * Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) detected during screening.
  * History of cardiac failure, significant/symptomatic bradycardia, Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome or any of the following:
  * Known risk to prolong the QT interval or induce Torsade's de Pointes.
  * Uncorrected hypomagnesemia or hypokalemia.
  * Systolic Blood Pressure (SBP) >160 mmHg or <90 mmHg.
  * Bradycardia (heart rate <50 at rest), by ECG or pulse.
  * On screening, inability to determine the QTcF interval on the ECG (i.e.: unreadable or not interpretable) or QTcF >450 screening ECG (based on a mean of 3 ECGs).
* History of hypersensitivity to ribociclib or any of its components.
* HIV-positive participants on combination antiretroviral therapy are ineligible. These participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Pregnant women are excluded from this study because the safety of ribociclib is not established in pregnant women. For this reason and because CDK4/6 agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of treatment, and for at least 3 months after the completion of treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Prior to study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential. All WOCBP must have a negative pregnancy test within 72 hours prior to receiving the first dose of the investigational agent(s). Registration may occur prior to this pregnancy test. If the pregnancy test is positive, the patient must not receive protocol treatment and must not be enrolled in the study. WOCBP is defined as follows: Any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or a bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea > 12 consecutive months, or women on hormone replacement therapy (HRT) with documented plasma follicle-stimulating hormone (FSH) level > 35 mIU/ml). Even women who are using oral, implanted, or injectable contraceptive hormones or mechanical products (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g. vasectomy), should be considered to be a WOCBP.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the study and for 8 weeks after study drug discontinuation. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential. Highly effective contraception methods include:

  * Total abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
  * In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment. Note: While oral contraceptives are allowed, they should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-12-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
ctDNA clearance | 12 Months
  tumor ctDNA response after 12 cycles of adjuvant ribociclib in combination with endocrine therapy vs endocrine therapy alone in patients with localized post-menopausal breast cancer and elevated ctDNA.

SECONDARY OUTCOMES:
Comparison of Adverse Events | 2 years
  compare the adverse effects, as assessed by CTCAE grading, in patients treated with endocrine therapy within 5 years versus those on endocrine therapy > 5 years
Number of participants who have a switch in endocrine therapy | 2 years
  determine how many patients have switch in endocrine therapy
Disease-free survival (DFS) | 2 years
  Disease-Free Survival (PFS) is defined as the time from randomization (or registration) to evidence of disease recurrence or death due to any cause. Participants alive without disease recurrence are censored at date of last evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Medford, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts

IPD SHARING:
Plan to Share IPD: No